CLINICAL TRIAL: NCT00478556
Title: Omnipaque Versus Gastroview as Oral Contrast for Abdominal and Pelvic CT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Michelle McNamara, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: F070208011; Omnipaque vs Gastroview Oral (Other: Department Name)
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Results first posted 2010-06-11 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: CT scan; oral contrast
MeSH Terms: interventions — Iohexol; Diatrizoate Meglumine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Gastroview
  Interventions: Drug: Gastroview
- 2 (Experimental): Omnipaque
  Interventions: Drug: Omnipaque

INTERVENTIONS:
Drug: Omnipaque — Oral CT contrast
  Other Names: Iohexol
  Arms: 2
Drug: Gastroview — Oral CT contrast
  Other Names: diatrizoate meglumine and diatrizoate sodium solution USP
  Arms: 1

SUMMARY:
Patients who are scheduled by their health care provider for routine computed tomography (CT) scan will be asked to participate in this study. The primary purpose is to determine if there is a difference in patient preference for Omnipaque versus Gastroview as oral contrast for abdominal pelvic CT. A secondary objective is to evaluate if there is significant difference in bowel opacification for the two agents.

DETAILED DESCRIPTION:
Participants must be scheduled for a CT scan prior to enrollment in this study. Informed consent will be obtained from patients acceptable to be included in the study. It will be noted if there is a history of gastrointestinal surgery and if the patient is nauseated before the contrast is administered.

Patients will be randomized to receive either a standardized dilution of Gastroview or Omnipaque orally. The two agents will be prepared to have nearly equivalent iodine concentration. No flavoring agent (ie Crystal Light) will be added. The plan is to mix the agents per manufacturer recommendation as follows:

Omnipaque 350 26cc in 974 cc of water (9.0g iodine) Gastroview 25cc in 1000cc of water (9.17g iodine)

The time the patients start and stop consuming the contrast as well as the volume taken and time from first drink to start of the scan will be recorded by a blinded investigator. Patients will be asked to drink 900cc. Technical staff will report any side effects or complications observed.

After completion of the CT scan, patients will fill in a survey rating the taste of the agent on a 5 point scale, and will be asked to report any side effects. Planned rating scale is as follows:

* 2=Dislike very much
* 1=Dislike moderately 0=Neither like nor dislike

  * 1=Like moderately
  * 2=Like very much

A taste test between the two agents will then be administered by a blinded investigator. Patients will be given 30 cc of each agent. The order in which the agents are administered will be randomized. Patients will be asked to rate preference, if any, for either agent on a 3 point scale. Potential bias related to which agent was administered for the CT will analyzed from the data.

Planned rating scale is as follows:

* 1- A is better 0 -no difference

  * 1- B is better

Patients will be contacted by telephone the day after the CT to assess for any delayed side effects such as diarrhea, constipation, and abdominal cramping experienced in the 24 hours following.

Bowel opacification will be rated by 2 body imagers blinded to the agent the patient received. Degree of opacification of the stomach, duodenum, jejunum, and ileum will be rated on a 4 point scale. If contrast has reached the colon, ascending, transverse, descending and sigmoid will be similarly evaluated. Four point rating scale is as follows:

0= absent opacification

1. minimal (<25% of analyzed segments opacified)
2. good (>25 % and < 75% of analyzed segments opacified)
3. excellent (> 75% of analyzed segments opacified)

Description of tests/procedures to be performed. Patients will undergo contrast enhanced abdominal pelvis CT as ordered by the referring clinician. Patients will be randomized to either dilute Omnipaque or dilute Gastroview for oral contrast. Both agents will be in a concentration of 9 mg of iodine/ml, and a volume of 900 cc.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 19 years of age scheduled for outpatient contrast enhanced abdominal pelvic CT at The Kirklin Clinic in Birmingham Alabama as part of clinical care with the patient's provider will be screened for eligibility.

Exclusion Criteria:

* Not competent to give consent.
* Pregnant.
* Known allergy to either of the contrast agents.
* Loss of sense of taste or smell.
* Contraindication to oral administration such as aspiration risk.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle McNamara, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Kirklin Clinic, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients will be randomized to receive either a standardized dilution of Gastroview or Omnipaque orally. The two agents will be prepared to have nearly equivalent iodine concentration.
Groups:
- Gastroview Group: Patients will be given oral Gastroview (contrast) prior to Computerized Tomography (CT).
- Omnipaque Group: Patients ill be given oral Omnipaque (contrast) prior to Computerized Tomography (CT).
Period: Overall Study
Arm/Group | Gastroview Group | Omnipaque Group
Started | 151 | 149
Completed | 151 | 149
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gastroview: Oral Gastroview prior to CT
- Omnipaque: Oral Omnipaque prior to CT
- Total: Total of all reporting groups
Arm/Group | Gastroview | Omnipaque | Total
Number analyzed (Participants) | 151 | 149 | 300
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 111 | 96 | 207
  >=65 years | 40 | 53 | 93
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (15) | 57 (15) | 57 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 56 | 116
  Male | 91 | 93 | 184
Region of Enrollment [Number; unit: participants]
  United States | 151 | 149 | 300

OUTCOME MEASURES:

1. Primary Outcome: Preferred Contrast Agent
Description: The primary outcome variable is the taste test when subjects will be asked which preparation they prefer. Possible answers include Onmipaque, Gastroview or neither.
Time Frame: 1 Day
Population: Analysis was per protocol
Measure: Number; unit: participants
Arm/Group | Gastroview | Omnipaque
Number analyzed (Participants) | 151 | 149
participants
  Prefer Gastroview | 25 | 29
  Prefer Omnipaque | 117 | 116
  No Preference | 9 | 4
Statistical Analysis 1: Comparison: Gastroview vs Omnipaque; All individuals tasted both preparations and indicated preference. A binomial test of proportion was done to see if these values differed from 50%; Test type: Superiority or Other; p < 0.001, Binomial test of proportion; tested if values were different from 50%; difference in proportions = 62

2. Secondary Outcome: Bowel Opacification Score
Description: The bowel opacification score was calculated by adding values for stomach, duodenum, jejunum and ileum for each patient. They were averaged across two doctors who read the studies. Scores can range from 0 (no opacification) to 3 (excellent) for each segment and from 0 to 12 for bowel opacification score.
Time Frame: Collected day of study
Population: per protocol - all patients had usable data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gastroview | Omnipaque
Number analyzed (Participants) | 151 | 149
units on a scale | 8.57 (1.96) | 8.85 (1.71)
Statistical Analysis 1: Comparison: Gastroview vs Omnipaque; Wilcoxon Rank Sum test was used to assess differences in bowel opacification score between the two groups; Test type: Superiority or Other; p = 0.270, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Arm/Group | Gastroview | Omnipaque
Serious Adverse Events (participants affected / at risk) | 0/151 | 0/149
Other Adverse Events (participants affected / at risk) | 0/151 | 0/149

LIMITATIONS AND CAVEATS:
Study was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No